CLINICAL TRIAL: NCT06862258
Title: Laparoscopic Vessel Sparing Descent of Intra-abdominal Testis: A Quasi-experimental Study.
Brief Title: Shehata Technique in the Treatment of Intra-abdominal Testis
Acronym: INP2024/063
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Pediatrics, Mexico (Other Government)
Responsible Party: Principal Investigator, Jose Francisco Gonzalez-Zamora, Clinical Professor, National Institute of Pediatrics, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INP 2024/063
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cryptorchidism
Keywords: Cryptorchidism; Shehata technique; intra-abdominal testis; Vessel Intact Laparoscopic Orchiopexy; testis atrophy
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intra-abdominal testis (Experimental): This single-arm quasi-experimental study involves subjects aged 6 months to 7 years with intra-abdominal cryptorchidism confirmed by laparoscopy. The subjects will be non-syndromic and may present with unilateral or bilateral cryptorchidism.
  In the case of a short testicular pedicle, participants will undergo laparoscopic testicular descent while preserving the testicular vessels. A two-stage descent will be performed using the elongation and delayed descent technique (Shehata).
  Six months post-operation, testicular atrophy (assessed for safety) and the position of the testis within the scrotum (assessed for efficacy) will be evaluated through ultrasonography and clinical examination. Each subject will serve as their own control by comparing outcomes before and after the intervention
  Interventions: Procedure: Shehata technique

INTERVENTIONS:
Procedure: Shehata technique — For patients whose intra-abdominal testicle cannot easily reach the contralateral internal inguinal ring due to a short testicular pedicle, the Shehata procedure will be performed. This technique involves a two-stage laparoscopic orchidopexy that preserves the testicular vessels. In the first stage, the intra-abdominal testicle is fixed above the contralateral iliac crest using prolene vascular suture. Twelve weeks later, a second procedure is performed to position the testicle lower. This approach ensures the preservation of the testicular vessels, vas deferens, and overall circulation.

SUMMARY:
This study focuses on children diagnosed with intra-abdominal cryptorchidism, a condition in which the testicle remains lodged in the abdomen instead of descending to the scrotum. The scrotum is the anatomical area where testicles should reside to maintain their viability and future reproductive function. Treating this condition typically requires one or two surgeries to relocate the testicle to the scrotum while preserving its vital structures, including the vas deferens, veins, and arteries that supply it with blood. In some cases, these structures are long enough to allow for a single surgery, which is referred to as the VILO technique. However, in other cases, the structures may be too short, making it necessary to perform two operations. In the first operation, the testicle is detached and moved to the opposite side of the abdomen while preserving its vital structures. This procedure aims to allow the artery, vein, and vas deferens to elongate over the next 12 weeks with the patient's movement. After this period, a second surgery can safely descend the testicle into the scrotum. This protocol specifically includes children with intra-abdominal testicles who will undergo one of two testicular vessel-preserving techniques: the Shehata technique or the VILO technique. If, during the first laparoscopic surgery, it is determined that the testicle is long enough to be descended safely, the VILO technique will be used to complete the procedure in a single surgery. If the length is insufficient, the Shehata technique will necessitate two surgeries as outlined above. The aim of this scientific research protocol is to prospectively document all clinical and intraoperative characteristics, along with the clinical and ultrasound postoperative evolution of your son, including several months after the final surgery. This study's objective is to evaluate both techniques for successfully relocating the testicle to the scrotum and to prevent any potential damage to the testicle during surge

DETAILED DESCRIPTION:
BACKGROUND AND STUDY AIMS Cryptorchidism, defined as the absence of one or both testicles from the scrotum, is the most common congenital genital anomaly identified at birth. The standard surgical treatment-orchiopexy-involves repositioning the testicle within the scrotal sac. Approximately 30% of cases involve "non-palpable testicles," which necessitate diagnostic laparoscopy as the preferred method for both diagnosis and treatment. A procedure is considered effective and safe when the testicle is successfully relocated to the scrotum without atrophy.

The most challenging form of cryptorchidism occurs when testicles are intra-abdominal with short testicular vessels, precluding primary descent. In these cases, the Fowler-Stephens technique has been developed; it involves dividing the testicular vessels to permit descent during a second surgical stage. However, this method is not without complications, with testicular atrophy being one of the most common adverse outcomes.

To address these issues, the Shehata technique was introduced in 2008, demonstrating a 100% success and safety rate in achieving scrotal descent without testicular atrophy. This impressive outcome relies on an intraoperative maneuver that assesses the vascular pedicle length, thereby guiding the choice of procedure (VILO vs. Shehata). Nonetheless, there is currently insufficient evidence to fully validate the significance of this maneuver. Therefore, the objectives of this study are to evaluate the safety and efficacy of the Shehata and VILO laparoscopic techniques for the descent of intra-abdominal testicles.

Who can participate? All patients from 6 months to 7 years of age, with intra-abdominal cryptorchidism confirmed by laparoscopy, non-syndromic, unilateral or bilateral What does the study involve? Patients will undergo a laparoscopic descent with preservation of testicular vessels, either a primary descent (VILO) or by means of the elongation and delayed descent technique (Shehata). Six months after surgery, testicular atrophy (safety) and intrascrotal placement (efficacy) will be determined by ultrasound and clinical examination, with the same subject being monitored before and after the intervention.

Where is the study run from? Instituto Nacional de Pediatría (México) When is the study starting and how long is it expected to run for? February 2025 to December 2025 Who is funding the study? Instituto Nacional de Pediatría (México) Who is the main contact? Silvio Carmona. Silviodocmor@hotmail.com STUDY DESIGN Study design: Quasi-experimental study Primary study design: Interventional Secondary study design: Quasi-Experimental Approach Study setting(s): Hospital Study type: Safety, Efficacy

Participant information sheet Study hypothesis

* The VILO technique will be effective and safe, with a success rate of over 90% and less than 5% testicular atrophy.
* The Shehata technique will be effective and safe, with a success rate of over 90% and less than 5% testicular atrophy.

Ethics approval(s) Approved: Dec 10 dic 2025, by Research Committee and Research Ethics Committee of the Instituto Nacional de Pediatria Number of Registry: 2024/063

Condition: Intrascrotal relocation of the intra-abdominal testicles is essential to improve the future fertility of patients,.

Intervention: Patients will be recruited from the surgical outpatient clinic with a diagnosis of cryptorchidism involving a non-palpable testicle. After a medical evaluation by an attending physician confirming the clinical presentation of a "non-palpable testicle," these patients will be invited to participate in the study. The parents of the participants will be informed about the patient's diagnosis, the available diagnostic and therapeutic options, and the necessary follow-up. The study protocol will include: a complete blood count, coagulation times, and a preoperative inguino-scrotal ultrasound .

The intraoperative measurement of the vascular pedicle length will determine whether the VILO or Shehata technique is employed.

VILO Group:

For patients whose intra-abdominal testicle reaches the contralateral internal inguinal ring without difficulty-and when, with the aid of a second laparoscopic clamp, the vascular pedicle and vas deferens can be elevated to contact the anterior abdominal wall , a primary descent will be performed.

Shehata Group:

For testicles that, despite gentle and extensive mobilization, require an attempt to lift the mesentery until it contacts the abdominal wall, if the resulting length is insufficient, a staged laparoscopic orchiopexy preserving the testicular vessel described by will be performed. This procedure involves contralateral fixation of the intra-abdominal testicle above the contralateral iliac crest using a vascular prolene suture, thereby preserving the testicular vessels as well as the vas deferens and its circulation. The procedure is then concluded with the closure of the laparoscopic incisions, and the patient is transferred to recovery.

Subsequently, a follow-up is scheduled at 12 weeks, preceded by an abdominal Doppler ultrasound to document the testicle's position and characteristics before the second surgical stage. During this second laparoscopic stage, once the testicle is located, it is freed from its fixation to the abdominal wall, and the final elongation of the vascular pedicle is documented using the same maneuver described by Shehata . The testicle is then descended through an ipsilateral paravesical neotract until it is externalized via an incision in the mid-third of the scrotum, where it is secured with two prolene sutures to the scrotal dartos.

Follow-Up Protocol:

• First Consultation (7-10 days postoperatively): Assessment of the healing of the laparoscopic incisions and, for those who underwent scrotal orchiopexy, the scrotal incision.

• Second Consultation (12-13 weeks postoperatively): Evaluation of the preliminary clinical outcomes regarding testicular position, and exclusion of postoperative complications such as inguinal hernia, umbilical hernia, and testicular atrophy. An inguino-scrotal ultrasound will also be performed to determine gonadal size and to re-measure both inguinal orifices.

• Third Consultation (6 months postoperatively): Clinical review, including a Doppler ultrasound evaluation to measure testicular volume, dimensions, and to assess for any abdominal wall defects.

• Fourth Consultation (12 months postoperatively): Clinical review, including a Doppler ultrasound evaluation to measure testicular volume, dimensions, and to assess for any abdominal wall defects.

• Annual Follow-Up: Color Doppler ultrasound examinations with testicular measurements and clinical evaluations.

Primary outcome measure Efficacy will be considered achieved if the corrected testicle remains in the lower or middle portion of the scrotum.

Safety will be determined by the preservation of more than 75% of the initial volume as calculated by ultrasound, maintenance of normal vascularity, or as assessed by direct measurements at the time of descent into the scrotum.

Secondary outcome measures Testicles that are positioned in the high or upper scrotum, those with a reduction in testicular volume to less than 75% of the original, or those with abnormalities on color Doppler will be considered as failed corrections.

The overall study start date is 01/01/2025 The overall study end date is 06/01/2027

Eligibility Participant type(s) Patient Age group 6 meses a 7 años de edad Sex Both Target number of participants 30 Participant inclusion criteria

* Patients with non-syndromic intra-abdominal cryptorchidism confirmed by laparoscopy.
* Patients whose parents or guardians sign an informed consent form for their inclusion.
* Patients from Mexico City or areas close to the city who can attend follow-up Participant exclusion criteria
* Patients with other concomitant genital abnormalities (e.g. hypospadias) Recruitment start date 02/25/2025 Recruitment end date 01/01/2026

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-syndromic intra-abdominal cryptorchidism confirmed by laparoscopy.
* Patients whose parents or guardians sign an informed consent form for their inclusion.
* Patients from Mexico City or areas close to the city who can attend follow-up

Exclusion Criteria:

* Patients with other concomitant genital abnormalities (e.g. hypospadias)

Ages: 6 Months to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Cryptorchidism in a male disease
Enrollment: 30 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Retraction | Basal, 12 weeks and 6 months
  Palpable testicle in the middle or lower third of the scrotum. Measuring scale: dichotomous: present/absent Number of measurements: 3 Measurement tool: Clinical review

SECONDARY OUTCOMES:
Testicular atrophy | Basal, 12 weeks and 6 months
  Measuring scale: dichotomous: present/absent Number of measurements: 3
  Measurement tool:
  The volume of both testicles in mm3 calculated by USG Doppler. Testicular atrophy is present if there is a difference of more than 25% in volume when comparing a healthy testicle with the affected one. Additionally, if the volume of the operated testicle decreases by more than 50% during monitoring, this also indicates testicular atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Carmona-Librado, MD, Principal Investigator — Instituto Nacional de Pediatria
Locations (1):
- Instituto Nacional de Pediatría, Mexico City, Coyoacan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The clinical data of the patients will be shared, taking care not to provide information that would allow them to be identified
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be available in March 2025 for 4 years.
Access Criteria: The IPD will be shared with the Institutional Research Committees and national regulatory authorities that require it, and, where appropriate, the journal's editorial committee to which the publication is requested. The information will be shared upon written request from the authorities mentioned above.
URL: https://www.pediatria.gob.mx/interna/ense_repositorio.html

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT06862258/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT06862258/ICF_001.pdf